CLINICAL TRIAL: NCT05236712
Title: Pilot Clinical Trial for a Mobile Health Intervention to Support Healthful Dietary Choices in Older Person
Brief Title: Mobile Health Intervention to Support Healthful Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Oleg Zaslavsky, Associate Professor: Biobehavioral Nursing & Health Informatics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00012842; K23AG059912-01A1 (NIH)
Record Dates: First submitted 2022-01-19; First posted 2022-02-11 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile health (Experimental): Participants will receive access to a mobile app installed on their device and will be asked to use the app at least once a week
  Interventions: Behavioral: Mobile app
- Usual care (No Intervention): Participants will receive information on public online resources

INTERVENTIONS:
Behavioral: Mobile app — The app sends reminder 'push' notifications to complete weekly surveys. The survey is a series of questions about foods and drinks participants had in the last week. Once the weekly survey is completed the app generates a personalized weekly report showing foods we encourage participants to eat more of, eat less of, or keep eating the same amount of. The app will also show menu recommendations for breakfast, lunch, dinner, and snacks that will help participants to eat healthier. Finally, the app also has a feature that allows chatting with the research team by sending and receiving in-app texts.
  Arms: Mobile health

SUMMARY:
This will be a pilot clinical trial to evaluate preliminary efficacy of a newly designed mobile intervention designed to support healthy eating in old people. The main scientific premise of this project is that mobile approaches are feasible for behavioral and metabolic improvements in the population of people 65+ with mild-to-moderate frailty. Specific Aim of this project is to describe feasibility, acceptability and initial efficacy of the newly designed mobile intervention in a pilot RCT. The pilot RCT, comparing usual care to usual care plus mobile intervention, will provide data on the sensitivity of outcome measures and estimated effect size to inform a larger RCT. Primary outcomes for the pilot RCT will include change in adherence to Mediterranean diet (MedD) score, change in insulin sensitivity measures, feasibility and acceptability. Secondary outcomes include MedD knowledge, self-efficacy, outcome expectation, self-regulation, social support, platform use and anthropometric and functional measures.

ELIGIBILITY:
Inclusion Criteria:

Age 65+

Mild to moderate frailty

Suboptimal diet

-

Exclusion Criteria:

1. Dependence in activities of daily living
2. Memory Impairment
3. Hearing or visual impairment
4. Unusual dietary restrictions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Zaslavsky, PhD, MHA, RN, Principal Investigator — University of Washington
Locations (1):
- Univeristy of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Su Y, Wu KC, Chien SY, Naik A, Zaslavsky O. A Mobile Intervention Designed Specifically for Older Adults With Frailty to Support Healthy Eating: Pilot Randomized Controlled Trial. JMIR Form Res. 2023 Nov 15;7:e50870. doi: 10.2196/50870. PMID 37966877

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Health | Usual Care
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Health | Usual Care | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (4.8) | 70.0 (3.9) | 71.27 (4.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Mediterranean Diet (MED) Adherence Score at 3 Months
Description: Alternative MED (aMED) score will be calculated using the Food Frequency Questionnaire (FFQ). aMED scores range from 0 (nonadherence) to 9 (perfect adherence)
Time Frame: baseline, 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
score on a scale | 2.63 (2.0) | -0.29 (1.38)

2. Primary Outcome: Change From Baseline HOMA-IR Score at 3 Months
Description: Insulin resistance scores, homeostatic model (HOMA-IR) was calculated with the following formula: fasting plasma glucose (in mmol/L) X fasting plasma insulin (in lU/mL) divided by 22.5. Higher score indicates worse insulin resistance. Typically, a HOMA-IR value of less than 1 is considered normal, indicating low insulin resistance.
Time Frame: baseline, 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
score on a scale | -0.18 (0.72) | 0.1 (0.74)

3. Secondary Outcome: Change From Baseline Mediterranean Diet Knowledge Score at 3 Months
Description: MedD knowledge will be assessed using the Mediterranean Diet Nutrition Knowledge (MDNK) Questionnaire. The total scores range from 0 to 30. Higher score higher knowledge
Time Frame: baseline, 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
score on a scale | 2.0 (2.33) | -1.14 (1.95)

4. Secondary Outcome: Change From Baseline Positive Outcome Expectations Score at 3 Months
Description: Questionnaire, 7 items rated on a 5-point scale (strongly agree 5; strongly disagree 1). Higher score more positive outcome expectations. The total scale ranges from 7 to 35
Time Frame: baseline, 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
score on a scale | 1.5 (5.26) | 1.0 (3.74)

5. Secondary Outcome: Change From Baseline Negative Outcome Expectations Score at 3 Months
Description: Questionnaire, 6 items rated on a 5-point scale (strongly agree 5; strongly disagree 1). Higher score more negative outcome expectations. The total score ranges from 30 to 6
Time Frame: baseline, 3 month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
score on a scale | -3.25 (3.62) | -0.43 (1.9)

6. Secondary Outcome: Change From Baseline Self-regulation Score at 3 Months
Description: Questionnaire, 2 items rated on a 5-point scale (strongly agree 5; strongly disagree 1). Higher score more self-regulation. The total scale ranges from 10 to 2
Time Frame: baseline, 3 month
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
score on a scale | -0.13 (1.25) | -1.86 (3.13)

7. Secondary Outcome: Change From Baseline Self-Efficacy Score at 3 Months
Description: Visual analog scale (VAS), 6 items using a 10-point scale. Higher values more self-efficacy. The total score ranges from O to 60
Time Frame: baseline, 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
score on a scale | 1.75 (10.59) | -2.0 (10.21)

8. Secondary Outcome: Change From Baseline Social Support Score at 3 Months
Description: Questionnaire, 2 items rated on a 5-point scale (strongly agree 5; strongly disagree 1). Higher score more social support. The total score ranges from 10 to 2
Time Frame: baseline, 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
score on a scale | 1.5 (1.41) | -0.14 (2.19)

9. Secondary Outcome: Change From Baseline Physical Performance Measure at 3 Months
Description: Short Physical Performance Battery (SPPB) is a composite measure assessing walking speed, standing balance, and sit-to-stand performance. The three tests are summed to give a total score, with a maximum of 12 and minimum of 0. Higher score higher function
Time Frame: baseline, 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
score on a scale | 1.5 (1.2) | 0.14 (0.9)

10. Secondary Outcome: Change From Baseline BMI at 3 Months
Description: BMI in units
Time Frame: baseline, 3 month
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Mobile Health | Usual Care
Number analyzed (Participants) | 8 | 7
Kg/m^2 | -0.83 (0.95) | -0.16 (0.65)

ADVERSE EVENTS:
Time Frame: three months
Arm/Group | Mobile Health | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT05236712/Prot_SAP_000.pdf